CLINICAL TRIAL: NCT02415816
Title: Diffusion Weighted Magnetic Resonance Imaging in Pediatric Sarcomas
Brief Title: Diffusion Weighted Magnetic Resonance in Imaging Younger Patients With Newly Diagnosed Bone or Soft Tissue Sarcomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DWSARC; NCI-2015-00290 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2015-04-09; First posted 2015-04-14 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Sarcoma, Bone; Sarcoma, Soft Tissue; Osteosarcoma; Sarcoma, Ewing; Rhabdomyosarcoma; Non-rhabdomyosarcoma Soft-tissue Sarcoma
Keywords: Pediatric; Whole body DWI MRI
MeSH Terms: conditions — Osteosarcoma; Sarcoma; Sarcoma, Ewing; Rhabdomyosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): All patients who consent to participate in this protocol. They will have diffusion weighted magnetic resonance imaging performed at several time points.
  Interventions: Procedure: Diffusion Weighted Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Diffusion Weighted Magnetic Resonance Imaging — Diffusion weighted magnetic resonance imaging (DWI MRI) is a method that does not involve radiation and can be used to assess the primary tumor as well as to image the entire patient, from head to toe. Diffusion weighted MRI uses a strong motion probing gradient to detect the movement of water in tissue. Tissues that are composed of tightly packed cells, such as tumors, allow less water movement than tissues with loosely packed cells. As tumors respond to therapy they become necrotic and cells are less tightly packed. This change in water diffusivity can be quantitated using DWI. Therefore, DWI provides a non-invasive, non-ionizing, and quantitative method of assessing tumor response at a cellular level and does not depend on a change in tumor size
  Other Names: DWI-MRI

SUMMARY:
Children with sarcomas are routinely assessed with a variety of imaging techniques that involve the use of ionizing radiation. These include computed tomography (CT), nuclear bone scan, and positron emission tomography-CT (PET-CT). Pediatric sarcoma patients undergo many imaging studies at the time of diagnosis, during therapy and for years following completion of therapy. Because children are in a stage of rapid growth, their tissues and organs are more susceptible to the harmful effects of ionizing radiation than are adults. Furthermore, compared to adults, children have a longer life expectancy and, therefore, a longer period of time in which to develop the adverse sequelae of radiation exposure, such as the development of second malignancies.

Alternative experimental methods of measuring tumor response will be compared to current standard of care measures to determine if the experimental method is equivalent to methods currently being used. Investigators wish to determine if they can reduce patient's exposure to the harmful effects of ionizing radiation by replacing imaging studies that use radiation with whole body diffusion weighted magnetic resonance imaging (DW-MRI) which does not use any radiation. They also want to know if DW-MRI measurements of the tumor can tell how well the tumor is responding to therapy. There have been studies in adults with cancer that have shown that DW-MRI provides useful information about how tumors are responding to therapy. There have only been very small studies of DW-MRI in children with tumors in the body. Therefore, the role of DW-MRI in pediatric sarcoma patients is not yet known and it is still experimental. This study might give us important information that could help us treat other children with bone or soft tissue sarcomas in the future.

DETAILED DESCRIPTION:
Whole body (WB) and primary tumor diffusion weighted imaging (DWI) will be performed at baseline in all subjects. Additional DW-MRIs will be done up to 3 times during treatment at the same time as routine MRI examinations are scheduled. Follow-up primary tumor DWI MRI examinations will be performed at time points determined by the participant's therapeutic treatment protocol. Follow-up primary tumor DWI examinations will be performed until completion of local control (surgical resection or completion of radiation therapy). All examinations will be performed on 1.5T Siemens magnetic resonance (MR) scanners unless there is a clinical indication for 3T imaging.

Because investigators will correlate imaging parameters with patient outcome, participants will be followed until they are discharged to the After Completion of Therapy Clinic or until they have tumor progression or recurrence or develop a second malignancy or death, whichever comes first.

PRIMARY OBJECTIVES:

* To estimate the proportion of pediatric sarcoma patients whose bone/bone marrow and soft-tissue metastasis status are correctly staged by whole body diffusion weighted MRI (WB DWI) at the time of diagnosis by comparing it to clinical stage.
* To determine the correlation between changes in primary pediatric sarcoma 18F-fluorodeoxyglucose positron emission tomography (FDG PET) maximum standardized uptake values (SUVmax) and average DWI apparent diffusion coefficient (ADC) values from baseline (pre-treatment) to just prior to local control.

OTHER PRESPECIFIED OBJECTIVES:

* To estimate the sensitivity, specificity, accuracy, and negative and positive predictive values of WB DWI, PET-CT and PET-CT + bone scan for detecting sites of metastatic tumor in pediatric sarcomas using biopsy or clinical follow-up (including imaging studies and clinical information) as the reference standards.
* To compare the ability of WB MRI, PET-CT and PET-CT + bone scan to detect all sites of metastases in pediatric sarcoma patients using biopsy and clinical judgment as the reference standards.
* To examine the associations of DWI ADC values of primary tumors at diagnosis and treatment protocol driven time points during therapy with tumor histology, tumor grade, RECIST response, % tumor necrosis, FDG SUVmax and patient outcome.
* To compare whole body DWI to conventional T1W and STIR whole body MRI for the detection of nodal, bone/bone marrow, soft-tissue or lung metastases among pediatric bone and soft-tissue sarcoma patients using biopsy and clinical judgment as the reference standards.
* To investigate the value of a variety of quantitative parameters obtained from software analysis of the primary tumor, such as; histogram kurtosis, range, peak, shifts in peak, or tumor heterogeneity.

ELIGIBILITY:
Inclusion Criteria:

* All St Jude patients with a known or suspected, newly diagnosed bone or soft-tissue sarcoma who will be treated on or as per disease specific protocols.
* Study subjects will have undergone or are scheduled for PET-CT and/or bone scan within about 2 weeks of the WB and primary tumor DWI MRI.
* No limit on age or gender
* Informed consent or assent signed by study subject or parent/guardian according to institutional guidelines.
* Patients should not have begun therapy, or, needed research imaging can be performed within 2-5 days of starting therapy.

Exclusion Criteria:

* Subject has a tumor that will undergo upfront resection
* Subject is unable or unwilling to follow study requirements, including signed consent or assent
* Subject is hospitalized in the intensive care unit.
* Subject does not meet institutional MRI safety screening requirements.
* Subject has undergone primary tumor resection prior to arrival at St. Jude.
* Subjects who require sedation for WB MRI will be excluded if they have:

  * An acute cardiopulmonary process including, but not limited to, croup, reactive airways disease, pneumonia, clinical or radiological evidence of pericardial effusion or other cardiopulmonary disease.
  * Vomiting within 24 hours of the MRI or substantial nausea that may preclude sedation as determined by the anesthesiologist or certified registered nurse anesthetist.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2015-06-05 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with pediatric sarcomas whose bone/bone marrow and soft-tissue metastasis status is correctly staged with whole body DWI MRI | Baseline, at time of diagnosis (day 0 within about 5 days)
  To allow for blinding, reading of scan images will be delayed at least 2 months and up to 6 months following scan.
  Proportion of participants whose bone/bone marrow and soft-tissue metastases were detected with whole body DWI MRI
The primary tumor DWI ADC and FDG PET SUVmax values at baseline and protocol driven time points up until local control | Baseline, at time of diagnosis (day 0 within about 5 days) to local control (up to 18 weeks)
  The primary tumor DWI ADC (in mm^2/sec) and FDG PET SUVmax (unitless) values at baseline and protocol driven time points up until local control.
  Local control is defined as surgical resection or initiation of radiation therapy.
  To allow for blinding, reading of scan images will be delayed at least 2 months and up to 6 months following scan.

OTHER OUTCOMES:
The number of metastatic lesions detected and not detected with whole body DWI MRI, PET-CT alone and PET-CT + bone scan at the time of diagnosis of a pediatric sarcoma | Baseline, at time of diagnosis (day 0 within about 5 days)
  The number of metastatic lesions detected and not detected with whole body DWI MRI, PET-CT alone and PET-CT + bone scan by using biopsy or clinical follow-up as the reference standards. Metastatic sites will be reported in groups by region (bone/bone marrow, lymph nodes, lung and soft-tissue) and all groups together.
  To allow for blinding, reading of scan images will be delayed at least 2 months and up to 6 months following scan.
The proportion of WB DWI MRIs, PET-CTs and PET-CT + bone scans that correctly identify sites of metastatic disease in patients with newly diagnosed sarcoma. | Baseline, at diagnosis (day 0 within about 5 days)
  The proportion of DWI MRI scans , PET-CTs and PET-CT + bone scan that correctly identify bone/bone marrow, nodal, lung and soft-tissue metastases in pediatric sarcoma patients at the time of diagnosis.
  To allow for blinding, reading of scan images will be delayed at least 2 months and up to 6 months following scan.
Primary tumor ADC values for each tumor histology group (osteosarcoma, Ewing sarcoma, non-rhabdomyosarcoma soft-tissue sarcoma and rhabdomyosarcoma (RMS) | Baseline, at diagnosis (day 0 within about 5 days) and at protocol driven time points up to 18 weeks (time of local control).
  To allow for blinding, reading of scan images will be delayed at least 2 months and up to 6 months following scan.
Primary tumor ADC values for low vs intermediate vs high grade tumors | Baseline, at diagnosis (day 0 within about 5 days) and at protocol driven time points up to 18 weeks (time of local control).
  To allow for blinding, reading of scan images will be delayed at least 2 months and up to 6 months following scan.
Primary tumor ADC values for tumors grouped by % necrosis in increments of 10% or 20% (i.e. 10%, 20% etc or 20%, 40% etc, whichever is most relevant) | Baseline, at diagnosis (day 0 within about 5 days) and at protocol driven time points up to 18 weeks (time of local control).
  To allow for blinding, reading of scan images will be delayed at least 2 months and up to 6 months following scan.
Primary tumor ADC values for RECIST response groups (complete remission, partial remission, stable disease, progressive disease) | Baseline, at diagnosis (day 0 within about 5 days) and at protocol driven time points up to 18 weeks (time of local control).
  To allow for blinding, reading of scan images will be delayed at least 2 months and up to 6 months following scan.
Primary tumor ADC values for FDG SUVmax values | Baseline, at diagnosis (day 0 within about 5 days) and at protocol driven time points up to 18 weeks (time of local control).
  To allow for blinding, reading of scan images will be delayed at least 2 months and up to 6 months following scan.
Event free survival) | Baseline, at diagnosis (day 0 within about 5 days) and at protocol driven time points up to 5 years after the end of therapy
  Event free survival is defined as the time between end of therapy and tumor progression/recurrence, development of a second malignancy or death, whichever comes first.
Overall survival | Baseline, at diagnosis (day 0 within about 5 days) up to 6 years after starting cancer therapy
  Overall survival is defined as the percentage of participants still alive at the end of follow-up after starting cancer therapy.
The proportion of WB DWI, T1W and STIR MRIs that correctly identify all sites of metastatic disease in patients with newly diagnosed pediatric sarcoma. | Baseline, at diagnosis (day 0 within 7±2 days)
  The proportion of WB DWI, T1W and STIR MRIs that correctly identify metastatic disease grouped by site (bone/bone marrow, lymph node, lung and soft-tissue) as well as all sites together.
  To allow for blinding, reading of scan images will be delayed at least 2 months and up to 6 months following scan.

CONTACTS AND LOCATIONS:
Overall Officials: Mary E. McCarville, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols